CLINICAL TRIAL: NCT00099788
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Multinational, Clinical Trial to Evaluate the Efficacy and Safety of Ranolazine vs Placebo in Patients With Non-ST Segment Elevation Acute Coronary Syndromes
Brief Title: Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST Elevation Acute Coronary Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Philip Sager, Vice President, Clinical Research, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT 3036; MERLIN TIMI 36
Record Dates: First submitted 2004-12-21; First posted 2004-12-21 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Myocardial Ischemia
Keywords: Acute Coronary Syndrome; Myocardial Infarction; Heart Attack; Angina; Chest pain; Ischemia; Non-ST Elevation Acute Coronary Syndrome
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome; Myocardial Infarction; Angina Pectoris; Chest Pain; Ischemia | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ranolazine
  Interventions: Drug: Ranolazine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — IV to oral transition.
  Other Names: Ranexa
  Arms: 1
Drug: Placebo — IV to oral transition.
  Arms: 2

SUMMARY:
MERLIN-TIMI 36 is a multi-national, double-blind, randomized, placebo-controlled, parallel-group clinical trial designed to evaluate the efficacy and safety of ranolazine during acute and long-term treatment in approximately 5,500 patients with non-ST elevation acute coronary syndromes (ACS) treated with standard therapy. The primary efficacy endpoint in MERLIN-TIMI 36 is time to first occurrence of any element of the composite of cardiovascular death, myocardial infarction or recurrent ischemia in patients with non-ST elevation ACS receiving standard therapy. The study also evaluates the safety of long-term treatment with ranolazine compared to placebo.

DETAILED DESCRIPTION:
Morrow DA, Scirica BM, Karwatowska-Prokopczuk E, Skene A, McCabe CH, Braunwald E; MERLIN-TIMI 36 Investigators. Evaluation of a novel anti-ischemic agent in acute coronary syndromes: design and rationale for the Metabolic Efficiency with Ranolazine for Less Ischemia in Non-ST-elevation acute coronary syndromes (MERLIN)-TIMI 36 trial. Am Heart J. 2006 Jun;151(6):1186.e1-9.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with non-ST elevation acute coronary syndrome
* Ischemic symptoms (more than or equal to 5 minutes) at rest within 48 hours of study entry
* At least one additional risk factor (e.g., elevated cardiac enzymes, ST-depression, diabetes)

Exclusion Criteria:

* Persistent acute ST-segment elevation
* Successful revascularization during the qualifying hospitalization, prior to study entry
* Acute pulmonary edema, hypotension, or evidence of cardiogenic shock
* Clinically significant liver disease
* End stage kidney disease requiring dialysis
* Concomitant use of drugs known to prolong the QT interval, or any digitalis drugs
* Use at study entry of drugs that are strong inhibitors of cytochrome P450 3A4
* Pregnant or lactating women, or women of child bearing potential not using an acceptable form of birth control

Additional study entry criteria will be evaluated during initial screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6560 (Actual)
Dates: Start 2004-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of any element of the composite of cardiovascular death, myocardial infarction or recurrent ischemia through the end of the follow-up in non-ST elevation ACS. | First occurrence

SECONDARY OUTCOMES:
Composite of cardiovascular death, myocardial infarction, or severe recurrent ischemia. Safety of long-term treatment with ranolazine compared to placebo; safety endpoints are death from any cause and symptomatic documented arrhythmia. | First occurence

CONTACTS AND LOCATIONS:
Overall Officials: David A Morrow, MD, Principal Investigator — The TIMI Study Group
Locations (1):
- The TIMI Study Group, Boston, Massachusetts, United States

REFERENCES:
- [Background] Morrow DA, Scirica BM, Karwatowska-Prokopczuk E, Skene A, McCabe CH, Braunwald E; MERLIN-TIMI 36 Investigators. Evaluation of a novel anti-ischemic agent in acute coronary syndromes: design and rationale for the Metabolic Efficiency with Ranolazine for Less Ischemia in Non-ST-elevation acute coronary syndromes (MERLIN)-TIMI 36 trial. Am Heart J. 2006 Jun;151(6):1186.e1-9. doi: 10.1016/j.ahj.2006.01.004. PMID 16781216
- [Derived] Zelniker TA, Morrow DA, Scirica BM, Furtado JD, Guo J, Mozaffarian D, Sabatine MS, O'Donoghue ML. Plasma Omega-3 Fatty Acids and the Risk of Cardiovascular Events in Patients After an Acute Coronary Syndrome in MERLIN-TIMI 36. J Am Heart Assoc. 2021 Apr 20;10(8):e017401. doi: 10.1161/JAHA.120.017401. Epub 2021 Apr 12. PMID 33840228
- [Derived] Gutierrez JA, Karwatowska-Prokopczuk E, Murphy SA, Belardinelli L, Farzaneh-Far R, Walker G, Morrow DA, Scirica BM. Effects of Ranolazine in Patients With Chronic Angina in Patients With and Without Percutaneous Coronary Intervention for Acute Coronary Syndrome: Observations From the MERLIN-TIMI 36 Trial. Clin Cardiol. 2015 Aug;38(8):469-75. doi: 10.1002/clc.22425. Epub 2015 Jun 8. PMID 26059896
- [Derived] Scirica BM, Belardinelli L, Chaitman BR, Waks JW, Volo S, Karwatowska-Prokopczuk E, Murphy SA, Cheng ML, Braunwald E, Morrow DA. Effect of ranolazine on atrial fibrillation in patients with non-ST elevation acute coronary syndromes: observations from the MERLIN-TIMI 36 trial. Europace. 2015 Jan;17(1):32-7. doi: 10.1093/europace/euu217. Epub 2014 Sep 10. PMID 25210025
- [Derived] Nieminen T, Scirica BM, Pegler JR, Tavares C, Pagotto VP, Kanas AF, Sobrado MF, Nearing BD, Umez-Eronini AA, Morrow DA, Belardinelli L, Verrier RL. Relation of T-wave alternans to mortality and nonsustained ventricular tachycardia in patients with non-ST-segment elevation acute coronary syndrome from the MERLIN-TIMI 36 trial of ranolazine versus placebo. Am J Cardiol. 2014 Jul 1;114(1):17-23. doi: 10.1016/j.amjcard.2014.03.056. Epub 2014 Apr 16. PMID 24852915
- [Derived] O'Malley RG, Bonaca MP, Scirica BM, Murphy SA, Jarolim P, Sabatine MS, Braunwald E, Morrow DA. Prognostic performance of multiple biomarkers in patients with non-ST-segment elevation acute coronary syndrome: analysis from the MERLIN-TIMI 36 trial (Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST-Elevation Acute Coronary Syndromes-Thrombolysis In Myocardial Infarction 36). J Am Coll Cardiol. 2014 Apr 29;63(16):1644-53. doi: 10.1016/j.jacc.2013.12.034. Epub 2014 Feb 13. PMID 24530676
- [Derived] Rhee JW, Wiviott SD, Scirica BM, Gibson CM, Murphy SA, Bonaca MP, Morrow DA, Mega JL. Clinical features, use of evidence-based therapies, and cardiovascular outcomes among patients with chronic kidney disease following non-ST-elevation acute coronary syndrome. Clin Cardiol. 2014 Jun;37(6):350-6. doi: 10.1002/clc.22253. Epub 2014 Jan 30. PMID 24481910
- [Derived] Scirica BM, Braunwald E, Belardinelli L, Hedgepeth CM, Spinar J, Wang W, Qin J, Karwatowska-Prokopczuk E, Verheugt FW, Morrow DA. Relationship between nonsustained ventricular tachycardia after non-ST-elevation acute coronary syndrome and sudden cardiac death: observations from the metabolic efficiency with ranolazine for less ischemia in non-ST-elevation acute coronary syndrome-thrombolysis in myocardial infarction 36 (MERLIN-TIMI 36) randomized controlled trial. Circulation. 2010 Aug 3;122(5):455-62. doi: 10.1161/CIRCULATIONAHA.110.937136. Epub 2010 Jul 19. PMID 20644019
- [Derived] Mega JL, Hochman JS, Scirica BM, Murphy SA, Sloan S, McCabe CH, Merlini P, Morrow DA. Clinical features and outcomes of women with unstable ischemic heart disease: observations from metabolic efficiency with ranolazine for less ischemia in non-ST-elevation acute coronary syndromes-thrombolysis in myocardial infarction 36 (MERLIN-TIMI 36). Circulation. 2010 Apr 27;121(16):1809-17. doi: 10.1161/CIRCULATIONAHA.109.897231. Epub 2010 Apr 12. PMID 20385930
- [Derived] Chisholm JW, Goldfine AB, Dhalla AK, Braunwald E, Morrow DA, Karwatowska-Prokopczuk E, Belardinelli L. Effect of ranolazine on A1C and glucose levels in hyperglycemic patients with non-ST elevation acute coronary syndrome. Diabetes Care. 2010 Jun;33(6):1163-8. doi: 10.2337/dc09-2334. Epub 2010 Mar 31. PMID 20357382
- [Derived] Morrow DA, Scirica BM, Sabatine MS, de Lemos JA, Murphy SA, Jarolim P, Theroux P, Bode C, Braunwald E. B-type natriuretic peptide and the effect of ranolazine in patients with non-ST-segment elevation acute coronary syndromes: observations from the MERLIN-TIMI 36 (Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST Elevation Acute Coronary-Thrombolysis In Myocardial Infarction 36) trial. J Am Coll Cardiol. 2010 Mar 23;55(12):1189-1196. doi: 10.1016/j.jacc.2009.09.068. PMID 20298924
- [Derived] Wilson SR, Scirica BM, Braunwald E, Murphy SA, Karwatowska-Prokopczuk E, Buros JL, Chaitman BR, Morrow DA. Efficacy of ranolazine in patients with chronic angina observations from the randomized, double-blind, placebo-controlled MERLIN-TIMI (Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST-Segment Elevation Acute Coronary Syndromes) 36 Trial. J Am Coll Cardiol. 2009 Apr 28;53(17):1510-6. doi: 10.1016/j.jacc.2009.01.037. PMID 19389561
- [Derived] Scirica BM, Morrow DA, Budaj A, Dalby AJ, Mohanavelu S, Qin J, Aroesty J, Hedgepeth CM, Stone PH, Braunwald E. Ischemia detected on continuous electrocardiography after acute coronary syndrome: observations from the MERLIN-TIMI 36 (Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST-Elevation Acute Coronary Syndrome-Thrombolysis In Myocardial Infarction 36) trial. J Am Coll Cardiol. 2009 Apr 21;53(16):1411-21. doi: 10.1016/j.jacc.2008.12.053. PMID 19371824
- [Derived] Morrow DA, Scirica BM, Chaitman BR, McGuire DK, Murphy SA, Karwatowska-Prokopczuk E, McCabe CH, Braunwald E; MERLIN-TIMI 36 Investigators. Evaluation of the glycometabolic effects of ranolazine in patients with and without diabetes mellitus in the MERLIN-TIMI 36 randomized controlled trial. Circulation. 2009 Apr 21;119(15):2032-9. doi: 10.1161/CIRCULATIONAHA.107.763912. Epub 2009 Apr 6. PMID 19349325
- [Derived] Morrow DA, Scirica BM, Karwatowska-Prokopczuk E, Murphy SA, Budaj A, Varshavsky S, Wolff AA, Skene A, McCabe CH, Braunwald E; MERLIN-TIMI 36 Trial Investigators. Effects of ranolazine on recurrent cardiovascular events in patients with non-ST-elevation acute coronary syndromes: the MERLIN-TIMI 36 randomized trial. JAMA. 2007 Apr 25;297(16):1775-83. doi: 10.1001/jama.297.16.1775. PMID 17456819
- See also: Related Info — http://www.timi.org